CLINICAL TRIAL: NCT01961947
Title: Phase 3 Study of ASP7374 -Approved Egg-derived Vaccine Controlled, Double-blind, Parallel Group Study in Adults ≥20 and <65 Years of Age-
Brief Title: Study of ASP7374, Cell-culture-derived Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMN Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7374-CL-0102
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Influenza; Vaccine
Keywords: ASP7374; Approved egg-derived vaccine; Prevention of seasonal influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP7374 group (Experimental)
  Interventions: Biological: ASP7374
- TIV group (Active Comparator)
  Interventions: Biological: approved egg-derived TIV

INTERVENTIONS:
Biological: ASP7374 — subcutaneous
  Arms: ASP7374 group
Biological: approved egg-derived TIV — subcutaneous
  Other Names: Influenza HA vaccine "SEIKEN"
  Arms: TIV group

SUMMARY:
The purpose of this study is to compare immunogenicity and safety of ASP7374 (cell-culture derived influenza vaccine) with those of approved egg-derived trivalent inactivated vaccine (TIV) in adults ≥20 and <65 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or medically stable, as judged on the basis of history and concurrent diseases.
* Subject understands procedure of the protocol and is willing to comply with the protocol.
* Written informed consent has been obtained.

Exclusion Criteria:

* Scheduled to receive another vaccine during the study.
* Received influenza HA vaccine within 180 days prior to screening.
* Received or scheduled to receive a live vaccine within 28 days prior to vaccination with the study vaccine, and received or scheduled to receive an inactivated vaccine or a toxoid within 7 days prior to vaccination with the study vaccine.
* Diagnosis of immune deficit in the past, has a family member (within the third degree of kinship) with a diagnosis of congenital immunodeficiency syndrome.
* Received one of the following medications or treatment prior to vaccination with the study vaccine.
* Received one of the following medications or treatment prior to vaccination with the study vaccine: Interferon formulation, Drugs which affect the immune system, corticosteroids, G-CSF, M-CSF, Human immunoglobulin products, Blood products, Blood transfusion
* History of anaphylactic shock or an allergic reaction such as generalized eruption due to food (including chicken, poultry, foodstuffs derived from chicken, et al.) or drug (including vaccines) allergies, fever ≥39.0°C within 2 days after the previous vaccination (influenza vaccine and others)
* History of seizures, except for febrile seizures in childhood

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
seroconversion rate of hemagglutination inhibition (HI) antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
geometric mean titer (GMT) of HI antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B

SECONDARY OUTCOMES:
seroprotection rate of HI antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
GMT ratio of HI antibody titer (Day 29/Day 1) | Day1 and Day 29
  evaluated for A/H1N1, A/H3N2, and B
seroconversion rate of neutralizing antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
seroprotection of neutralizing antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
GMT of neutralizing antibody titer | Day 29
  evaluated for A/H1N1, A/H3N2, and B
GMT ratio of neutralizing antibody titer (Day 29/Day 1) | Day 1 and Day 29
  evaluated for A/H1N1, A/H3N2, and B
Local and systemic reactions associated with the vaccination | Day 1 through Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Principal Investigator — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Kanto
  - Kyushu